CLINICAL TRIAL: NCT06837532
Title: Ultrasound Guided Versus Surgical Rectus Sheath Block Versus Local Anesthesia Infiltration for Postoperative Analgesia in Patients Undergoing Total Abdominal Hysterectomy: A Randomized Trial
Brief Title: Ultrasound Guided Versus Surgical Rectus Sheath Block Versus Local Anesthesia Infiltration for Postoperative Analgesia in Patients Undergoing Total Abdominal Hysterectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah Ahmed, Lecturer of Anesthesia, Intensive care, and pain management, Faculty of Medicine, Ain Shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU R23/2025
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Ultrasound; Surgical; Rectus Sheath Block; Local Anesthesia Infiltration; Postoperative Analgesia; Total Abdominal Hysterectomy
MeSH Terms: interventions — Bupivacaine; Anesthesia, Local

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasound-guided rectus sheath block group (Experimental): Patients will receive ultrasound-guided rectus sheath block (20 ml bupivacaine 0.25%) bilaterally at the end of surgery.
  Interventions: Drug: Ultrasound-guided rectus sheath block
- Surgical rectus sheath block group (Experimental): Patients will receive a surgical rectus sheath block (20 ml bupivacaine 0.25%) bilaterally at the time of closure.
  Interventions: Drug: Surgical rectus sheath block
- Local anesthesia infiltration group (Experimental): Patients will receive local anesthesia infiltration at the end of surgery.
  Interventions: Drug: Local anesthesia infiltration

INTERVENTIONS:
Drug: Ultrasound-guided rectus sheath block — Patients will receive ultrasound-guided rectus sheath block (20 ml bupivacaine 0.25%) bilaterally at the end of surgery.
  Other Names: Bupivacaine
  Arms: Ultrasound-guided rectus sheath block group
Drug: Surgical rectus sheath block — Patients will receive a surgical rectus sheath block (20 ml bupivacaine 0.25%) bilaterally at the time of closure.
  Other Names: Bupivacaine
  Arms: Surgical rectus sheath block group
Drug: Local anesthesia infiltration — Patients will receive local anesthesia infiltration at the end of surgery.
  Other Names: Bupivacaine
  Arms: Local anesthesia infiltration group

SUMMARY:
The aim of this work is to compare the efficacy and safety of the effectiveness and safety of ultrasound-guided surgical rectus sheath block and local anesthetic infiltration for postoperative analgesia in patients undergoing total abdominal hysterectomy.

DETAILED DESCRIPTION:
Total abdominal hysterectomy (TAH) is a commonly performed major surgical procedure that results in substantial postoperative pain and discomfort.

Local anesthetic infiltration (LAI) at the end of surgery is one of the most common technique employed in laparotomies for postoperative analgesia.

Rectus sheath block (RSB) has been used as a part of multimodal analgesia, especially when neuraxial techniques are unsuitable.The RSB was used to achieve peri-operative relaxation of the anterior abdominal wall.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years old.
* American Society of Anesthesiologists (ASA) physical status I - II.
* Patients scheduled for elective total abdominal hysterectomy under general anesthesia.

Exclusion Criteria:

* Hepatic, renal or cardiac disease.
* Any known allergy to local anesthetic.
* Physical or mental conditions which may vaguely measure postoperative pain following surgery.
* History of chronic use of analgesic as nonsteroidal anti-inflammatory drugs (NSAIDs) or central nervous system (CNS) depressants as antiepileptic, and bleeding disorders.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women scheduled for elective total abdominal hysterectomy
Enrollment: 90 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the Visual Analogue Scale (VAS)> 3 to be repeated after 30 min if pain persists until the VAS < 4.

SECONDARY OUTCOMES:
Heart rate | Till the end of surgery (Up to 4 hours)
  Heart rate will be recorded preoperatively, before the block is performed, and every 15 minutes until the end of the surgery.
Mean arterial pressure | Till the end of surgery (Up to 4 hours)
  Mean arterial pressure will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.
Time to the first request for the rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of morphine administrated).
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at PACU, 2, 4, 6, 12, 18, and 24h postoperatively.
Degree of patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as hematoma, nerve damage or neuropathy, bradycardia, hypotension, nausea, vomiting, pruritis, urinary retention, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.